CLINICAL TRIAL: NCT01196065
Title: A Single Center, Open-label, Fixed Sequence, Two-period Study to Investigate the Effect of Memantine on Pharmacokinetics, Safety and Tolerability of RO5313534 After Single Dose Administration in Healthy Volunteers and the Effect of RO5313534 on Safety and Tolerability of Steady State Memantine
Brief Title: A Study of the Effect of Memantine on Pharmacokinetics, Safety and Tolerability of Single Dose RO5313534 in Healthy Volunteers, and the Effect of RO5313534 on Safety and Tolerability of Steady State Memantine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP25180; 2010-020080-20
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Memantine

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO5313534; Drug: memantine

INTERVENTIONS:
Drug: RO5313534 — single oral dose
Drug: memantine — multiple doses to steady state

SUMMARY:
This open-label, fixed sequence, two-period study will assess the effect of memantine on the pharmacokinetics, safety and tolerability of a single oral dose of RO5313534 and the effect of RO5313534 on safety and tolerability of steady-state memantine. Healthy volunteers will receive a single oral dose of RO5313534 on Day 1 of Treatment Period 1 (3 days). After a washout period of 5-21 days, oral memantine will be administered on Days 1-21 of Treatment Period 2 and a single dose of RO5313534 on Day 19. There will be a follow-up of 3-4 weeks after the last dose. Anticipated time on study for each volunteer is up to 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, 18 to 45 years of age inclusive
* Body mass index (BMI) 18-30 kg/m2
* Male subjects must agree to use a barrier method of contraception from first dosing until the end of the study
* Female subjects must be either surgically sterile or agree to use two forms of contraception until the end of the study
* Non-smoker for at least 6 months

Exclusion Criteria:

* Clinically significant history or detection during medical interview/physical examiation of any disease or condition that is capable of altering the absorption. metabolism or elimination of drugs, or would constitute a risk factor when taking the study drug
* History of drug addiction or alcohol abuse
* Any confirmed significant allergic reaction to any drug, or multiple allergies in the judgement of the investigator
* Positive serology to hepatitis B or hepatitis C or Human Immunodeficiency Viruses (HIV type 1 and 2) at screening
* Pregnant or lactating women
* Participation in an investigational drug or device study within the last 3 months prior to first dose

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Study Completion 2010-11

PRIMARY OUTCOMES:
Effect of multiple-dose memantine on single-dose pharmacokinetics of RO5313534 and of RO5313534 on steady-state pharmacokinetics of memantine | Days 16-21

SECONDARY OUTCOMES:
Effect of multiple-dose memantine on safety and tolerability of single-dose RO5313534 | up to 14 weeks
Safety and tolerability of memantine alone and in combination with a single dose of RO5313534 | up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rennes, France